CLINICAL TRIAL: NCT03199482
Title: A Comparative Evaluation of Effect of Dexamethazone on Postendodontic Pain and Success of Inferior Alveolar Nerve Block in Mandibular Molars With Symptomatic Irreversible Pulpitis
Brief Title: Effect of Pretreatment Dexamethazone on Pain and Success of Nerve Block
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Mohamed Safei Eldin Sayed, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: kinda
Record Dates: First submitted 2017-06-18; First posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: dexamethazone
Who Masked: Participant, Care Provider
Masking Description: investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Drug dexamethasone (Active Comparator): preoperative single dose of dexamethasone 0.5 mg oral tablet given to patients before starting of root canal treatment by 30 minutes.
  Interventions: Drug: Dexamethasone Oral Tablet
- Placebo (Placebo Comparator): Placebo will be administrated to patients before stating of root canal treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone Oral Tablet — single dose of tablet 0.5 mg dexamethasone given to patients before starting of root canal treatment by 30 minutes or placebo
  Arms: Drug dexamethasone
Drug: Placebo — Placebo will be administrated 30 minutes before start of root canal treatment
  Arms: Placebo

SUMMARY:
A Comparative Evaluation of the effect of pretreatment dexamethasone versus placebo on post-endodontic pain and success of inferior alveolar nerve block in Mandibular molars with symptomatic Irreversible Pulpitis: A Blinded Randomized Clinical Trial Therapeutic study

DETAILED DESCRIPTION:
Participants, Interventions and Outcome

Setting:

Patients are of the clinic of endodontics at the faculty of oral and dental medicine, Cairo University, Urban area, Cairo governorate, Egypt.

* The dental Unit is Adec 200 U.S.A.
* The x-ray Machine is ViVi, S.r.I, Italy
* The x-ray films are Kodac, speed D, size 2.
* The operators are master degree students in the department of Endodontics.
* No dental assistant
* Time: 2017-2016

Procedure steps:

1. Patients are asked to rate the pain level on numerical rating scale before the administration of drug to get the baseline record for the pain preoperatively.
2. Thirty minutes before the endodontic procedure,dexamethasone (0.5 mg) or a placebo will be administered.Root canal therapy in all cases was completed in a single visit.
3. After explanation of the treatment procedures (according to individual needs), the tooth will be anesthetized by an inferior alveolar nerve block (1.8 ml mepivacaine hydrochloride 2% 1: 100,000 epinephrine) using a side loading aspirating syringe and 27-gauge long needle.
4. At 15-minutes post injection, access cavity will be performed using round bur size 4 and endo-z bur and the pain is recorded .
5. Tooth is then isolated using rubber dam to prevent introduction of saliva and Bactria from the oral cavity.
6. Checking the patency of the canal with K- file size 10 taper 0.02, extirpation of pulp with H-file size 15 taper 0.02 with recording the pain.
7. Cleaning and shaping will be performed with a hybrid technique using hand K-files and rotary files for all teeth.
8. Irrigation will be performed with 2.5% NaOCl after each instrument in all cases. At the end of instrumentation, the final irrigation will made by saline.
9. After drying the canals with sterile paper points, they will be coated with AD-Seal sealer and obturated with gutta-percha using the lateral condensation technique.
10. The tooth will be then temporized by using cavit temporary filling and reduced from occlusion.
11. A rescue medication (ibuprofen) will be prescribed and the patients will be instructed to take it only if they experienced severe pain postoperatively. If rescue medication will be taken within the 48 hours after the treatment, then the patient will be excluded from the study.

Patients will be asked to make a mark on the point that represents level of perceived pain. (before the commencement of any treatment [baseline score]; at access and pulp extirpation, immediately after treatment completion; and 6, 12, 24, and 48 hours after the commencement of treatment). All subjects will be recalled after 2 days to return the pain diary and for a clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in good health with no systemic disease (American Society of Anesthesiologists Class II)
2. Patients having symptomatic irreversible pulpitis in one of their mandibular molars
3. Age range is between 20 and 50 years
4. Patients who can understand the categorical tool (points) for measurement
5. Patients able to sign informed consent

Exclusion Criteria:

1. Patients with positive percussion test
2. Patients having history of necrosis with or without apical pathosis
3. Patients have sinus tract or fistula extraoral or intraoral
4. Patients having active pain in more than one molar
5. Patients who had taken analgesics in the 12 hours preceding the preparation.
6. Complicating systemic disease
7. Subjects with allergies and hypersensitivity to or unable to take dexamethasone
8. Teeth with grade 2 or 3 mobility

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2017-07-12 (Estimated); Primary Completion 2017-10-12 (Estimated); Study Completion 2018-07-07 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 48 hours
  Numerical rating scale

SECONDARY OUTCOMES:
success of inferior alveolar nerve block | 2 hours
  Numerical rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Manar Hamouda, Professor, Study Director — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo, Manyal, Egypt

IPD SHARING:
Plan to Share IPD: No